CLINICAL TRIAL: NCT01301677
Title: Double-blind, Randomised, Active (Hydrocortisone) Controlled Study of the Effect of 10% w/v Strontium Chloride Hexahydrate on Ultraviolet B Radiation (UVR) Induced Signs of Inflammation (Erythema and Pain) in Healthy Volunteers
Brief Title: Ultra Violet B Radiation (UVR) Study of Strontium Chloride Hexahydrate Hydrocortisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X-pert Med GmbH (Industry)
Responsible Party: Ilka Rother, MD, X-pert Med GmbH
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: XPM-033
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Erythema; Pain
MeSH Terms: conditions — Erythema; Pain | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydrocortisone (Active Comparator)
  Interventions: Drug: Hydrocortisone
- 2PX+ (Experimental): strontium chloride hexahydrate in a penetration enhancing vehicle
  Interventions: Drug: 2PX+
- 2PX- (Experimental): strontium chloride hexahydrate without a penetration enhancing vehicle
  Interventions: Drug: 2PX-

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone liquid formulation
  Arms: Hydrocortisone
Drug: 2PX+ — strontium chloride hexahydrate in a penetration enhancing vehicle
  Arms: 2PX+
Drug: 2PX- — strontium chloride hexahydrate without a penetration enhancing vehicle
  Arms: 2PX-

SUMMARY:
Double blinded (subject and observer), randomised, active (hydrocortisone (HC)) controlled study of the effect of strontium chloride hexahydrate on ultraviolet B radiation (UVR) induced signs of inflammation (erythema and pain) in healthy volunteers.

DETAILED DESCRIPTION:
Subjects that signed the informed consent and are eligible to the study will be irradiated on the back to evaluate their individual minimal erythema dose (MED).

A training session (without study medication) will be performed in order to introduce subjects to the testing and rating procedures.

Subjects will come in within 28 days of screening to start the treatment period of the study.

For eligible subjects, three test areas oriented along the long axis of the back and different from the areas of MED determination will be defined for the evaluation of effects on pain and inflammation induced by UVR. The three areas will be irradiated with 2 MED. In addition, non-irradiated, not treated areas will serve as reference and training areas for the individual visits.

Topical treatments will be randomly assigned to the three test areas.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-mandated procedure
* Subjects in good health as determined by the Investigator
* Willing and able to comply with study requirements
* Age ≥ 18
* Fitzpatrick skin types I, II, or III
* Willing to avoid sun exposure, tanning lamps and use of any topical products on the test areas during the study
* Willing not to wash test areas during treatment period
* Willing to abstain from sauna, exposure to extreme cold or major physical activities during the treatment period of the study
* For females, subjects of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year) must be using appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner). Oral contraceptive medications are allowed in this study. Female subjects, who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) are also allowed for participation

Exclusion Criteria:

General

* Planned treatment or treatment with another investigational drug within 30 days prior to randomization.
* Subjects who are inmates of psychiatric wards, prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Pregnancy or lactation
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease.

Medical History

* Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma
* Known hypersensitivity or allergy (including photoallergy) to hydrocortisone, strontium chloride hexahydrate, glycofurol, dimethylsulphoxide (DMSO), ethanol, propylene glycol, glycerol, hypomellose, sodium edentate, sodium hydroxide, citric acid monohydrate and metagin
* History of photosensitivity disease
* Sunburn, excessive tan, uneven skin tones or blemishes of the test areas
* Pain conditions which might interfere with pain rating during the study, e.g. neuropathic pain
* Open wounds, infection, inflammation or other dermal diseases of the intended application areas
* ALT or AST ≥ 5 times the ULN
* Glomerulary filtration rate < 30 ml/min

Medication History

* Systemic or topical drugs that might affect responses to UVR or interfere with responses to IMP including corticosteroids, thiazides, tetracyclines and NSAIDs must be washed out with 5 times half-life time prior to randomization to treatment
* Drugs with potential dermatologic adverse events defined by the respective summary of product characteristics (e.g. tetracyclines, gyrase inhibitors) must be washed out with 5 times half-life time prior to randomization to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Degree of erythema | at 6 h, 12 h, 24 h, 36 h, 48 h post UVR

SECONDARY OUTCOMES:
Pain threshold (primary hyperalgesia to heat) | Sum of assessments at 6 h, 12 h, 24 h, 36 h, 48 h post UVR

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Rother, MD, Principal Investigator — X-pert Med GmbH
Locations (2):
- Germany (2):
  - X-pert Med GmbH, Gräfelfing, Bavaria
  - X-pert Med Gmbh, Jena, Thuringia